CLINICAL TRIAL: NCT07328542
Title: A Multi-center, Open-label, Single-arm 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Study of Testosterone Cypionate Injection in Hypogonadal Men
Brief Title: Ambulatory Blood Pressure Monitoring (ABPM) Study in Hypogonadal Men
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Azurity Pharmaceuticals (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ-01022-7300-002
Record Dates: First submitted 2026-01-07; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hypogonadism, Male
Keywords: Hypogonadal Men; Ambulatory Blood Pressure Monitoring (ABPM)
MeSH Terms: conditions — Eunuchism | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Testosterone Cypionate Injection (Experimental)
  Interventions: Drug: Testosterone Cypionate Injection 200 mg/mL

INTERVENTIONS:
Drug: Testosterone Cypionate Injection 200 mg/mL — Participants will receive Testosterone Cypionate Injection 200 mg/mL at established dose during the titration and treatment periods every two weeks (± 2 days) as a deep intramuscular injection in the gluteal muscle for 14-week study duration.

SUMMARY:
A Phase 4, multi-center, open-label, single-arm 24-hour Ambulatory Blood Pressure Monitoring (ABPM) study of Testosterone Cypionate Injection in Hypogonadal Men to assess change in 24-hour ambulatory blood pressure from Baseline to End of Treatment

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥18 to ≤75 years of age (inclusive) at time of enrollment.
* Body mass index (BMI) ≥17 kg/m^2 to < 40 mg^2.
* Willing and able to voluntarily provide written informed consent prior to initiation of screening or study-specific procedures.
* Able to understand and to follow the protocol requirements, restrictions, and instruction, in the Investigator's opinion
* Diagnosed with primary hypogonadism (congenital or acquired) or hypogonadotropic hypogonadism (congenital or acquired).
* Hypogonadal males (individual serum testosterone concentrations <350 ng/dL and mean serum testosterone concentrations <300 ng/dL, determined from at least two samples separated at least 48 hours apart and obtained between 6 AM and 10 AM local time).
* Testosterone therapy naïve or has discontinued current treatment and completed adequate washout of prior androgen therapy or any other therapy which causes significant change in serum androgen level i.e., clomiphene, anabolic steroids, compounded or over-the-counter androgenic steroid derivatives and dehydroepiandrosterone (45 days or 5 half-lives of the drug, whichever is longer, prior to collection of baseline serum testosterone samples). Washout must be completed prior to collection of baseline serum testosterone samples to determine study eligibility.
* An office blood pressure measurement <140 millimeters of mercury (mmHg) for SBP AND <90 mmHg for DBP.
* If the subject is on an antihypertensive regimen, he has been on stable dose for at least 4 weeks prior to study enrollment.
* If the subject is on glucocorticoids >7.5 mg prednisone equivalent per day (e.g., hydrocortisone 30 mg, methylprednisolone 6 mg, or dexamethasone 1.2 mg), he has been on stable dose for at least 4 weeks prior to study enrollment with no intention of changing dose for the duration of the study.
* Subjects with acceptable laboratory parameters

  1. Hematocrit ≤ Upper limit of normal (ULN)
  2. Hemoglobin ≤ 16 gm%
  3. Prolactin ≤ ULN
  4. PSA ≤ 4.0 ng/mL (PSA level between 1.5 to 4.0 ng/mL (both inclusive) for subject who is treated with 5-alpha reductase inhibitors (e.g., dutasteride, finasteride)
  5. HbA1c ≤ 9 %
  6. ALT ≤ 2.5 x ULN
  7. AST ≤ 2.5 x ULN
  8. Serum bilirubin ≤ 2.0 mg/dL
* No history of addiction to any recreational drug or drug dependence or alcohol abuse (including illicit steroid use) as per Investigator's judgement.
* Subject is not considering fathering a child or donating sperm during the study or for approximately 30 days after the last dose of study drug.
* Subject is not currently enrolled in another clinical study and will not enroll in another clinical study throughout the duration of the study.

Exclusion Criteria:

* Subjects with known hypersensitivity to study drug, including androgens, or product excipients.
* Subjects with abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or International Prostate Symptom Score (I-PSS) score > 19 points.
* Subjects with history of, or current or suspected, prostate or breast cancer.
* Subjects with history of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study enrollment except for diabetes, or renal disease
* Subject with history of fluid or electrolyte imbalance.
* Subject taking anticoagulant.
* Subjects with history of uncontrolled heart failure, stroke or myocardial infarction within the past 6 months.
* Subject with history of severe lower urinary tract symptoms in past 6 months.
* Subjects with history of diagnosed, severe, untreated, obstructive sleep apnea.
* Subjects working night shifts.
* Subjects performing strenuous manual labor or exercise while wearing the ABPM monitor.
* Subjects with chronic atrial fibrillation or any other chronic condition, which interferes with the ability to obtain precise ambulatory recordings.
* Subject with polycythemia.
* Subject with history of thrombophilia or venous thromboembolic events.
* Subject with positive serology for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Human Immunodeficiency Virus (HIV).
* Participation in any clinical study within 45 days or 5 half-lives of the drug before dosing of Investigational Product.
* Loss of ≥ 350 ml (1 unit) of blood within 30 days of enrollment in the study.
* Any other medical condition or serious inter current illness that, in the opinion of the Investigator, may make it undesirable for the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with changes in 24-hour average systolic ambulatory blood pressure | From Baseline to End of Treatment, up to Week 14 (Day 99)

SECONDARY OUTCOMES:
Number of participants with changes in 24-hour average diastolic ambulatory blood pressure | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in 24-hour average pulse pressure | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in 24-hour average heart rate | From Baseline to End of Treatment, up to Week 14 (Day 99)
Percent of participants taking new antihypertensive medications | From Baseline to End of Treatment, up to Week 14 (Day 99)
Percent of participants requiring increases in dose of antihypertensive medications from baseline | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in daytime average systolic blood pressure (SBP) | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in daytime average diastolic blood pressure (DBP) | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in daytime mean arterial pressure (MAP) | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in daytime average pulse pressure | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in daytime average heart rate | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in night time average systolic blood pressure (SBP) | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in night time average diastolic blood pressure (DBP) | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in night time mean arterial pressure (MAP) | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in night time average pulse pressure | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with changes in night time average heart rate | From Baseline to End of Treatment, up to Week 14 (Day 99)
Number of participants with drug-related adverse events | From Baseline to End of Treatment, up to Week 14 (Day 99)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Hillcrest Medical Research, LLC, DeLand, Florida
  - Integrity Clinical Research Center, Inc., Hialeah, Florida
  - AccuMed Research Associates, Garden City, New York
  - Aim Trials, Plano, Texas
  - Alpine Clinical Organization Inc., Clinton, Utah